CLINICAL TRIAL: NCT01588509
Title: An Open-label, Randomized Study to Estimate the Percent Change From Baseline in Lumbar Spine Bone Mineral Density After 3 Months of AMG 785 Administration in Postmenopausal Women With Low Bone Mineral Density Previously Treated With Alendronate
Brief Title: Transition From Alendronate to Romosozumab (AMG 785)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20110253
Record Dates: First submitted 2012-04-17; First posted 2012-05-01 (Estimated); Results first posted 2019-03-04 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Osteoporosis
Keywords: AMG 785, bone mineral density, alendronate
MeSH Terms: conditions — Osteoporosis | interventions — romosozumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Romosozumab 140 mg (Experimental): Participants received romosozumab 140 mg administered subcutaneously once a month for 3 months.
  Interventions: Drug: Romosozumab
- Romosozumab 210 mg (Experimental): Participants received romosozumab 210 mg administered subcutaneously once a month for 3 months.
  Interventions: Drug: Romosozumab

INTERVENTIONS:
Drug: Romosozumab — Administered by subcutaneous injection
  Other Names: AMG 785; EVENITY™

SUMMARY:
The purpose of this study is to estimate the percent change from baseline in lumbar spine bone mineral density (BMD) following multiple-dose administrations of romosozumab in postmenopausal women with low BMD previously treated with alendronate.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women, defined as no vaginal bleeding or spotting for ≥ 12 months
* Low bone mineral density at screening [defined by a bone mineral density (BMD) T-score ≤ -2.0 and ≥ -4.0 at the lumbar spine (L1 to L4; or BMD T-score of evaluable vertebrae), total hip, or femoral neck]
* Currently taking alendronate (70 mg weekly or equivalent) exclusively for ≥ 1 year with verbal agreement that the subject has taken ≥ 80% of their doses with good tolerance

Exclusion Criteria:

* History of vertebral fracture, or fragility fracture of the wrist, humerus, hip or pelvis after age 50; or recent bone fracture within 6 months prior to screening
* History of metabolic or bone disease such as Paget's disease, rheumatoid arthritis, osteomalacia, osteogenesis imperfecta, osteopetrosis, ankylosing spondylitis, Cushing's disease, hyperprolactinemia, and malabsorption syndrome
* Vitamin D deficiency (defined as 25-OH-VitD levels < 20 ng/mL)

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03-30 (Actual); Primary Completion 2012-11-21 (Actual); Study Completion 2012-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (9):
- United States (9):
  - Research Site, Tucson, Arizona
  - Research Site, Walnut Creek, California
  - Research Site, Gainesville, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Bethesda, Maryland
  - Research Site, Albuquerque, New Mexico
  - Research Site, West Haverstraw, New York
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Seattle, Washington

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 8 centers in the United States. The first participant enrolled on 30 March 2012 and the last participant enrolled on 21 August 2012.
Period: Overall Study
Arm/Group | Romosozumab 140 mg | Romosozumab 210 mg
Started | 30 | 30
Received Treatment | 30 | 30
Completed | 29 | 30
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Romosozumab 140 mg | Romosozumab 210 mg | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (7.5) | 66.7 (8.3) | 66.1 (7.8)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 14 | 15 | 29
  ≥ 65 years | 16 | 15 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 14 | 26
  Not Hispanic or Latino | 18 | 16 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Black (or African American) | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Other | 0 | 1 | 1
  White | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) at the Lumbar Spine
Description: Bone mineral density was assessed by dual energy X-ray absorptiometry (DXA) scans of the lumbar spine (L1-L4) and analyzed by a central imaging lab.
Time Frame: Baseline and day 85
Population: All participants who received study drug and with non-missing baseline and day 85 measurements.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 29 | 30
percent change | 2.13 (0.64) | 2.08 (0.63)
Statistical Analysis 1: Comparison: Romosozumab 140 mg; Test type: Superiority; p = 0.002, ANOVA; Percent Change from Baseline = 2.13, 90% CI 2-sided [1.05 to 3.20]
Statistical Analysis 2: Comparison: Romosozumab 210 mg; Test type: Superiority; p = 0.002, ANOVA; Percent Change from Baseline = 2.08, 90% CI 2-sided [1.02 to 3.14]

2. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) at the Femoral Neck
Description: Bone mineral density was assessed by dual energy X-ray absorptiometry (DXA) scans and analyzed by a central imaging lab.
Time Frame: Baseline and day 85
Population: All participants who received study drug and with non-missing baseline and day 85 measurements.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 29 | 30
percent change | 2.06 (0.59) | 1.92 (0.58)
Statistical Analysis 1: Comparison: Romosozumab 140 mg; Test type: Superiority; p < 0.001, ANOVA; Percent Change from Baseline = 2.06, 90% CI 2-sided [1.07 to 3.05]
Statistical Analysis 2: Comparison: Romosozumab 210 mg; Test type: Superiority; p = 0.002, ANOVA; Percent Change from Baseline = 1.92, 90% CI 2-sided [0.95 to 2.89]

3. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) at the Total Hip
Description: Bone mineral density was assessed by dual energy X-ray absorptiometry (DXA) scans and analyzed by a central imaging lab.
Time Frame: Baseline and day 85
Population: All participants who received study drug and with non-missing baseline and day 85 measurements.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 29 | 30
percent change | 1.38 (0.34) | 1.40 (0.34)
Statistical Analysis 1: Comparison: Romosozumab 140 mg; Test type: Superiority; p < 0.001, ANOVA; Percent Change from Baseline = 1.38, 90% CI 2-sided [0.81 to 1.95]
Statistical Analysis 2: Comparison: Romosozumab 210 mg; Test type: Superiority; p < 0.001, ANOVA; Percent Change from Baseline = 1.40, 90% CI 2-sided [0.84 to 1.96]

4. Secondary Outcome: Percent Change From Baseline in Serum Type-1 Aminoterminal Propeptide (P1NP)
Time Frame: Baseline and days 4, 15, 29, 43, 57, 71, and 85
Population: All participants who received study drug and with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 30 | 30
percent change
  Day 4 | 22.1263 (3.3852) | 30.4935 (4.9950)
  Day 15 | 140.9970 (15.1975) | 218.4994 (22.6148)
  Day 29 | 128.3936 (17.7834) | 221.9954 (23.3718)
  Day 43 | 164.1654 (17.7832) | 251.0495 (23.4572)
  Day 57: number analyzed (Participants) | 29 | 30
  Day 57 | 99.3682 (14.9155) | 168.7689 (17.1565)
  Day 71: number analyzed (Participants) | 28 | 30
  Day 71 | 127.4051 (14.8572) | 205.2619 (23.5171)
  Day 85: number analyzed (Participants) | 29 | 30
  Day 85 | 64.9103 (10.5005) | 142.5601 (20.3233)

5. Secondary Outcome: Percent Change From Baseline in Serum C-telopeptide (sCTX)
Time Frame: Baseline and days 4, 15, 29, 43, 57, 71, and 85
Population: All participants who received study drug and with available data at each time point
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 30 | 30
percent change
  Day 4 | -28.2149 (3.9352) | -14.8099 (4.6844)
  Day 15 | -28.9365 (4.6974) | -22.2800 (5.1854)
  Day 29 | 3.1008 (8.6448) | -1.8188 (7.4121)
  Day 43 | 3.4511 (8.9913) | 11.0131 (10.0244)
  Day 57: number analyzed (Participants) | 29 | 30
  Day 57 | 25.7433 (8.7440) | 35.7697 (13.5346)
  Day 71: number analyzed (Participants) | 28 | 30
  Day 71 | 28.4465 (11.7345) | 44.3802 (13.7159)
  Day 85: number analyzed (Participants) | 29 | 30
  Day 85 | 54.0549 (14.2140) | 61.1734 (13.9874)

6. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical trial participant.
  Laboratory value changes that required treatment or adjustment in current therapy were considered adverse events.
  A treatment-related adverse event (TRAE) was an adverse event assessed by the investigator as possibly related to the investigational product, indicated by a "yes" response to the question: Is there a reasonable possibility that the event may have been caused by the investigational product?
  A serious adverse event was defined as an adverse event that met at least 1 of the following serious criteria:
  * fatal,
  * life-threatening,
  * required in-patient hospitalization or prolongation of existing hospitalization,
  * resulted in persistent or significant disability/incapacity,
  * congenital anomaly/birth defect, and/or
  * other medically important serious event.
Time Frame: From first dose of study drug up to day 85
Population: All participants who received study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 30 | 30
Participants
  All adverse events | 14 | 15
  Serious adverse events | 0 | 0
  AE leading to discontinuation of study drug | 0 | 0
  AE leading to discontinuation from study | 0 | 0
  Fatal adverse events | 0 | 0
  Treatment-related adverse events | 3 | 4
  Treatment-related serious adverse events | 0 | 0
  TRAE leading to discontinuation of study drug | 0 | 0
  TRAE leading to discontinuation from study | 0 | 0
  Treatment-related fatal adverse events | 0 | 0

7. Secondary Outcome: Number of Participants Who Developed Anti-romosozumab Antibodies
Description: Two validated assays were used to detect the presence of anti-romosozumab antibodies. An electrochemiluminescent bridging immunoassay was used to detect binding antibodies (screening assay) and confirm antibodies (confirmatory assay) capable of binding romosozumab. Samples testing positive in the immunoassay were further tested in a competitive binding bioassay for neutralizing activity against romosozumab. If a sample was positive for binding antibodies and demonstrated neutralizing activity, the participant was defined as positive for neutralizing antibodies. Participants who developed anti-romosozumab antibodies were those with a negative result at baseline and a positive result at any time postbaseline.
Time Frame: Baseline and days 29, 57, and 85
Population: All participants who received study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 30 | 30
Participants
  Binding antibody positive | 2 | 2
  Neutralizing antibody positive | 0 | 0

8. Secondary Outcome: Mean Serum Concentration of Romosozumab
Time Frame: Days 4, 15, 29, 43, 57, 71 and 85
Population: All participants who received study drug with available data at each time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 30 | 30
ng/mL
  Day 4: number analyzed (Participants) | 22 | 26
  Day 4 | 15000 (6350) | 23200 (9730)
  Day 15: number analyzed (Participants) | 30 | 29
  Day 15 | 10500 (3540) | 18500 (6640)
  Day 29: number analyzed (Participants) | 30 | 29
  Day 29 | 3890 (2000) | 8200 (4470)
  Day 43 | 14300 (4280) | 22800 (9390)
  Day 57: number analyzed (Participants) | 29 | 30
  Day 57 | 5490 (2600) | 10700 (6380)
  Day 71: number analyzed (Participants) | 28 | 30
  Day 71 | 13700 (5000) | 22700 (10500)
  Day 85: number analyzed (Participants) | 29 | 30
  Day 85 | 5350 (3190) | 11600 (6850)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to day 85
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Romosozumab 140 mg | Romosozumab 210 mg
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 11/30 | 6/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Romosozumab 140 mg (N=30) | Romosozumab 210 mg (N=30)
Fatigue (General disorders) | 3 | 0
Injection site reaction (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.